CLINICAL TRIAL: NCT05347056
Title: The Effect of Vertebral Body Tethering on Lumbar Paraspinal Muscle Cross-Section Area, Lumbar Range of Motion and Trunk Muscle Strength in Adolescent Idiopathic Scoliosis
Brief Title: The Effect of Vertebral Body Tethering on Lumbar Paraspinal Muscle Cross-Section Area in Adolescent Idiopathic Scoliosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Esin Nur Taşdemir, MD, Istanbul University
Other Study IDs: ENTASDEMIR
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Idiopathic Scoliosis
Keywords: Scoliosis; Vertebral body tethering; Motion preservation; Multifidus; Magnetic resonance imaging
MeSH Terms: conditions — Scoliosis | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vertebral Body Tethering Group: Vertebral Body Tethering applied to the lumbar region, with or without fusion to the thoracic region
  Interventions: Diagnostic Test: Lumbar Spine Magnetic Resonance; Diagnostic Test: Isokinetic trunk flexion-extension trunk muscle strength and endurance test; Diagnostic Test: Lomber Region Range of motion assessment; Diagnostic Test: Radiograph; Behavioral: SRS 22
- Selective Thoracic Fusion Group: selective thoracic fusion was applied, no intervention was applied to the lumbar region
  Interventions: Diagnostic Test: Lumbar Spine Magnetic Resonance; Diagnostic Test: Isokinetic trunk flexion-extension trunk muscle strength and endurance test; Diagnostic Test: Lomber Region Range of motion assessment; Diagnostic Test: Radiograph; Behavioral: SRS 22

INTERVENTIONS:
Diagnostic Test: Lumbar Spine Magnetic Resonance — Metal artifact reduction sequence (mars), axial t2 sequence
Diagnostic Test: Isokinetic trunk flexion-extension trunk muscle strength and endurance test — To evaluate for trunk muscle strength and endurance angular velocity of 60 and 120°/s
  Other Names: Cybex
Diagnostic Test: Lomber Region Range of motion assessment — To evaluate for lomber region ROM with digital inclinometer
Diagnostic Test: Radiograph — spinal radiograph AP/Lateral
Behavioral: SRS 22 — SRS-22 Patient Questionnaire

SUMMARY:
We aimed to compare the paraspinal muscle cross-section area and functional results of anterior vertebral tethering and selective thoracic fusion surgery.

DETAILED DESCRIPTION:
Idiopathic scoliosis is a three-dimensional deformity of the spine. It is defined as the curvature of the spine of 10° or more detected radiologically in the coronal plane. In scoliosis, changes in axial rotation in the transverse plane and physiological curvatures in the sagittal plane (decrease or increase in kyphosis, lordosis) occur.

The incidence of scoliosis is 2-3%, but up to 10% of patients need surgical treatment. Knowing the long-term effects of posterior spinal fusion is currently the gold standard treatment because it gives good results in deformity improvement. However, fusion surgery has disadvantages such as loss of motion in the spine and long-term development of adjacent segment disease and disc degeneration. It has also been suggested that spinal fusion causes iatrogenic damage to the paraspinal muscles (especially the multifidus), which is of great importance in the alignment and movement of the spine due to the posterior approach during surgery.

As a result of damage to the lumbar multifidus muscles and the development of fatty degeneration, problems such as spinal sagittal alignment disorders and chronic low back pain can be seen. In addition, fatty degeneration and atrophy of the paraspinal muscles may lead to the development of adjacent segment disease in the segments under fusion in the long term.

In selective thoracic fusion, by protecting the mobile segments in the lumbar region, the range of motion is preserved and iatrogenic damage of the lumbar paraspinal muscles is prevented. After selective thoracic fusion (STF), some improvement occurs in the deformity in the lumbar region. However, the risk of insufficient improvement and progression of the curve in the unfused lumbar segments, especially in immature patients, should be considered.

Anterior vertebra body tethering is a surgical technique that has been used more frequently in recent years, which is thought to prevent functional complications caused by spinal fusion.With this method, which allows the growth of the spine to continue, there is no need for fusion when treating progressive curvature. Short-term radiological results of this surgical technique have been reported frequently in recent years, but the literature on functional results (spine flexibility, trunk endurance, etc.) is very limited.

In our study, we plan to evaluate the effects of AVT applied to the lumbar region on paraspinal muscle quality, trunk muscle strength and endurance, and trunk joint range of motion by evaluating patients who underwent selective thoracic fusion surgery and patients who underwent thoracic fusion + AVT to the lumbar region.

ELIGIBILITY:
Inclusion Criteria:

Males or females age 12 to 19 years old Diagnosis of idiopathic scoliosis At least 6 months have passed since surgical intervention Spina bifida occulta is permitted

Exclusion Criteria:

Pregnancy Prior spinal or chest surgery MRI abnormalities (including syrinx greater than 4mm, Chiari malformation, or tethered cord) Neuromuscular, thoracogenic, cardiogenic scoliosis, or any other non-idiopathic scoliosis Associated syndrome, including Marfan syndrome or neurofibromatosis

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: At least 6 months have passed since the surgical procedure, Patients followed in Istanbul Medical Faculty Department of Orthopedics and Traumatology Group 1: VBT applied Group 2: only selective thoracic fusion was applied
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2022-05-09 (Estimated); Primary Completion 2022-05-27 (Estimated); Study Completion 2022-06-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of VBT and STF group paraspinal muscles cross-section area | 6 months to 3 years after surgery
  The bilateral cross-sectional areas (CSA) of the multifidus (MF), erector spinae (ES) and psoas (P) muscles at all disc levels were measured by outlining the fascial boundary of the muscle
Comparison of pre-op and post-op paraspinal muscles cross-section area | 6 months to 3 years after surgery
  The bilateral cross-sectional areas (CSA) of the multifidus (MF), erector spinae (ES) and psoas (P)

SECONDARY OUTCOMES:
Investigation of Quality of Life in Adolescent Idiopathic Scoliosis | 6 months to 3 years after surgery
  Quality of life Scoliosis Research Society-22 (SRS-22) questionnaire
Comparison of VBT and STF group trunk muscle strenght and endurance | 6 months to 3 years after surgery
  Cybex Norm
Comparison VBT and STF group lomber range of motion | 6 months to 3 years after surgery
  Dual inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Esin Nur Taşdemir, MD, Principal Investigator — Istanbul Medicine Faculty Department of Sports Medicine

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Green DW, Lawhorne TW 3rd, Widmann RF, Kepler CK, Ahern C, Mintz DN, Rawlins BA, Burke SW, Boachie-Adjei O. Long-term magnetic resonance imaging follow-up demonstrates minimal transitional level lumbar disc degeneration after posterior spine fusion for adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2011 Nov 1;36(23):1948-54. doi: 10.1097/BRS.0b013e3181ff1ea9. PMID 21289549
- [Result] Pehlivanoglu T, Oltulu I, Erdag Y, Akturk UD, Korkmaz E, Yildirim E, Sarioglu E, Ofluoglu E, Aydogan M. Comparison of clinical and functional outcomes of vertebral body tethering to posterior spinal fusion in patients with adolescent idiopathic scoliosis and evaluation of quality of life: preliminary results. Spine Deform. 2021 Jul;9(4):1175-1182. doi: 10.1007/s43390-021-00323-5. Epub 2021 Mar 8. PMID 33683642
- [Result] Kim HJ, Yang JH, Chang DG, Suk SI, Suh SW, Nam Y, Kim SI, Song KS. Long-Term Influence of Paraspinal Muscle Quantity in Adolescent Idiopathic Scoliosis Following Deformity Correction by Posterior Approach. J Clin Med. 2021 Oct 19;10(20):4790. doi: 10.3390/jcm10204790. PMID 34682913
- [Result] Baroncini A, Trobisch PD, Berrer A, Kobbe P, Tingart M, Eschweiler J, Da Paz S, Migliorini F. Return to sport and daily life activities after vertebral body tethering for AIS: analysis of the sport activity questionnaire. Eur Spine J. 2021 Jul;30(7):1998-2006. doi: 10.1007/s00586-021-06768-6. Epub 2021 Feb 27. PMID 33638722